| Informed consent for participation in a health science research project. |
|---|
| Title of the research project: ASSESSMENT OF DIAPHRAGM FUNCTION. A METHOD STUDY AND A CLINICAL STUDY. |
| May 15. 2019. |
| Statement from the subject: |
| I have received written and oral information and I know enough about the purpose, method, advantages and disadvantages to agree to participate. |
| I understand that participation is voluntary and that I can always withdraw my consent without losing my current or future rights to treatment. |
| I give my consent to participate in the research project and have received a copy of this consent form and a copy of the written information about the project for my own use. |
| Subject's name: |
| Date Signature: |
| Do you want to be informed about the results of the research project and any consequences for you?: |
| Yes (set x) No (set x) |
| Declaration by the person providing the information: |
| I declare that the subject has received oral and written information about the experiment. |
| In my opinion, sufficient information has been provided for a decision to be made regarding participation in the trial. |
| The name of the person who submitted the information: |
| Date Signature: |